CLINICAL TRIAL: NCT02172521
Title: Effect of Spiriva® 18 Microgram on Health-related Quality of Life and Physical Functioning in Patients With COPD and Proven Hyperinflation
Brief Title: Effect of Spiriva® 18 Microgram on Health-related Quality of Life and Physical Functioning in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Proven Hyperinflation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.320
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD and proven hyperinflation: Patients with COPD and proven hyperinflation receiving tiotropium bromide 18 microgram
  Interventions: Drug: Tiotropium bromide

INTERVENTIONS:
Drug: Tiotropium bromide — Tiotropium bromide18 micrograms by oral inhalation (1 x daily) with the HandiHaler®
  Other Names: Spiriva®

SUMMARY:
* Primary objective of this observational study was to gain insights into the effects of therapy with Spiriva® (tiotropium bromide) 18 microgram on the health-related quality of life and physical functioning in patients with chronic obstructive pulmonary disease (COPD) and demonstrated hyperinflation.
* Secondary objective was to obtain safety data regarding adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with diagnosis of chronic obstructive pulmonary disease (COPD) with a thoracic gas volume (TGV) > = 120% as measured by body plethysmography
* Only patients who have not yet been treated with Spiriva® 18 micrograms can be included in the study.

Exclusion Criteria:

* Patients who presenting the general and specific contraindications mentioned in the Patient Information and Prescribing Information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1536 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline for assessment of the health-related euro quality of life 5 dimensions questionnaire (EQ-5D) time trade off (TTO) score | At baseline (visit 1) and after 4 weeks (visit 2)
Change from baseline for assessment of the health-related EQ-5D questionnaire linear rating scale | At baseline (visit 1) and after 4 weeks (visit 2)
Change from baseline for assessment of physical functioning in every day life (PF-10) | At baseline (visit 1) and after 4 weeks (visit 2)